CLINICAL TRIAL: NCT00152724
Title: Etude de la Reserve Vasomotrice Microcirculatoire cutanée
Brief Title: Mechanisms of Human Cutaneous Microcirculation in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CP96-04
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2007-03

CONDITIONS: Healthy Volunteers
Keywords: Physiology; Microcirculation; Laser-Doppler Flowmetry
MeSH Terms: interventions — Iontophoresis; Lidocaine, Prilocaine Drug Combination; Capsaicin; Aspirin; Clopidogrel; Celecoxib; Indomethacin; Acetylcholine; Nitroprusside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pressure strain system, iontophoresis
Drug: scopolamin
Drug: emla
Drug: capsaicin
Drug: aspirin
Drug: clopidogrel
Drug: celecoxib
Drug: indomethacin
Drug: acetylcholine
Drug: sodium nitroprusside
Drug: brethyllium
Device: general and local heating

SUMMARY:
Microvascular dysfunctions are critical events in several diseases including diabetes. This study will develop a methodology for microvascular investigation in human skin. The purpose of the study is to investigate the physiological response of the cutaneous microcirculation to physical, thermal, mechanical or chemical stimulations.

DETAILED DESCRIPTION:
This study has investigated various aspects of the physiology of the microcirculation in the past years and is still recruiting under parallel protocols of physiological investigations of the neurovascular control of the cutaneous microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with no clinical signs of, or risk factors for, vascular disease

Exclusion Criteria:

* Smokers, Pregnancy, Allergy,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 1996-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Amplitude of the vasomotor response to stimuli | 1 hour

SECONDARY OUTCOMES:
Kinetics of the vasomotor response to stimuli | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis SAUMET, MD - PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Laboratoire de Physiologie et Explorations Vasculaires - CHU Angers, Angers, France

REFERENCES:
- [Result] Tartas M, Durand S, Koitka A, Bouye P, Saumet JL, Abraham P. Anodal current intensities above 40 microA interfere with current-induced axon-reflex vasodilatation in human skin. J Vasc Res. 2004 May-Jun;41(3):261-7. doi: 10.1159/000078665. Epub 2004 May 19. PMID 15153776
- [Result] Durand S, Fromy B, Humeau A, Sigaudo-Roussel D, Saumet JL, Abraham P. Break excitation alone does not explain the delay and amplitude of anodal current-induced vasodilatation in human skin. J Physiol. 2002 Jul 15;542(Pt 2):549-57. doi: 10.1113/jphysiol.2002.022731. PMID 12122152
- [Result] Tartas M, Bouye P, Koitka A, Durand S, Gallois Y, Saumet JL, Abraham P. Early vasodilator response to anodal current application in human is not impaired by cyclooxygenase-2 blockade. Am J Physiol Heart Circ Physiol. 2005 Apr;288(4):H1668-73. doi: 10.1152/ajpheart.00415.2004. Epub 2004 Nov 24. PMID 15563538
- [Result] Durand S, Tartas M, Bouye P, Koitka A, Saumet JL, Abraham P. Prostaglandins participate in the late phase of the vascular response to acetylcholine iontophoresis in humans. J Physiol. 2004 Dec 15;561(Pt 3):811-9. doi: 10.1113/jphysiol.2004.069997. Epub 2004 Oct 21. PMID 15498811
- [Result] Durand S, Fromy B, Tartas M, Jardel A, Saumet JL, Abraham P. Prolonged aspirin inhibition of anodal vasodilation is not due to the trafficking delay of neural mediators. Am J Physiol Regul Integr Comp Physiol. 2003 Jul;285(1):R155-61. doi: 10.1152/ajpregu.00742.2002. PMID 12793996
- [Result] Durand S, Fromy B, Koitka A, Tartas M, Saumet JL, Abraham P. Oral single high-dose aspirin results in a long-lived inhibition of anodal current-induced vasodilatation. Br J Pharmacol. 2002 Oct;137(3):384-90. doi: 10.1038/sj.bjp.0704868. PMID 12237259
- [Result] Durand S, Fromy B, Bouye P, Saumet JL, Abraham P. Vasodilatation in response to repeated anodal current application in the human skin relies on aspirin-sensitive mechanisms. J Physiol. 2002 Apr 1;540(Pt 1):261-9. doi: 10.1113/jphysiol.2001.013364. PMID 11927685